CLINICAL TRIAL: NCT04146441
Title: Ultrasound-enhanced Uptake of Chemotherapy in Patients With Inoperable Pancreatic Ductal Adenocarcinoma - A Randomized Controlled Trial
Brief Title: Ultrasound-enhanced Uptake of Chemotherapy in Patients With Inoperable Pancreatic Ductal Adenocarcinoma
Acronym: PDAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 040376MH; 2019-001736-57 (EudraCT Number)
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Carcinoma, Pancreatic Ductal
Keywords: Contrast agent BR; SonoVue; Ultrasonic therapy; Microbubbles
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal | interventions — contrast agent BR1; Drug Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SonoVue (Experimental): SonoVue + chemotherapy
  Interventions: Combination Product: SonoVue; Drug: Chemotherapy
- control (Active Comparator): chemotherapy
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Combination Product: SonoVue — 1,0 ml SonoVue 8ul/ml dispersion is given 9 times at 3,5 minute intervals 9 times, a total dosage of 9 ml. The experimental treatment lasts for 31,5 minutes every treatment day. Administered by authorized site personnel only
  Arms: SonoVue
Drug: Chemotherapy — FOLFIRINOX Regime according to Norwegian national guidelines

SUMMARY:
Patients with inoperable pancreatic cancer have extremely poor prognosis with five year survival below 8% in Norway. Life-prolonging chemotherapy has very limited effect, but is the only therapeutic option for these patients. This tumor is characterized by poor uptake and chemoresistance. Toxic effects on healthy tissue restrict doses applied and maintenance of treatment intensity. This severely limits clinical outcome. Increasing the local uptake of chemotherapy has potential benefits for patients in connection to side effects, survival and possible cure. Treatment with Focused Ultrasound (FUS) combined with microbubbles (MBs) is proved promising to improve treatment response in animal and clinical trials. Ultrasound can induce biological effects deep inside the body without surgical intervention. This opens for local delivery of drugs at desired sites. FUS in combination with regular contrast MBs has been reported to influence the delivery of drugs to tumors.

In this trial FUS and MB will be applied to locally advanced pancreatic cancers shortly after the administration of conventional chemotherapy. Primary aim of the trial is to investigate whether the effect of the cytostatic drug, measured in tumor volume, can be increased.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically verified stage III or IV PDAC or medically inoperable stage IIB T3 PDAC
* eligible for 1st line treatment with FOLFIRINOX, Gemcitabine -nab Paclitaxel, or Gemcitabine monotherapy.
* ECOG 0 - 1

Exclusion Criteria:

* Known contraindications for SonoVue
* Hematological bleeding status before experimental treatment:
* Hb < 8g/dL, trc < 80 x10 superscr 9/l, APTT˃ 45s, INR ˃ 1,5
* Pregnancy

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Volume change of primary tumor | 8 weeks
  measured by segmented tumor volumes on Computed Tomography of primary PDAC tumor from before treatment (baseline) to after 1 cycle of treatment

SECONDARY OUTCOMES:
Number of down-staged tumors from stage III to stage II | 8 weeks
Number of down-staged tumors from stage III to stage II | 1 year
Rate of reported toxicity | 8 weeks
  Toxicity reported by patients during structured interview after treatment. Type of side effects and severity according to Common Toxicity Criteria (CTC)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Hofsli, md phd, Study Director — St. Olavs Hospital
Locations (1):
- Department of Radiology, St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification(text, tables, figures, and appendices). Interested researchers who provide a reasonable, sound proposal are encouraged to direct this to the first author.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Protocol can be shared beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a reasonable, sound proposals are encouraged to direct this to the first author at margrete.haram@stolav.no